CLINICAL TRIAL: NCT03463538
Title: A Randomised Control Trial of Arthroscopic Capsular Release Versus Hydrodilatation for Primary Adhesive Capsulitis of the Shoulder
Brief Title: Hydrodilatation Versus Arthroscopic Capsular Release for Frozen Shoulder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal Devon and Exeter NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1312873
Record Dates: First submitted 2018-02-28; First posted 2018-03-13 (Actual); Last update posted 2018-03-14 (Actual); Status verified 2018-03

CONDITIONS: Frozen Shoulder
MeSH Terms: conditions — Bursitis | interventions — Joint Capsule Release

STUDY DESIGN:
Intervention Model Description: randomised control trial between interventions
Who Masked: Outcomes Assessor
Masking Description: independent clinical reviewer of patients ROM and collection of outcome scores
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arthroscopic capsular release (Active Comparator): Surgical release performed under general anesthetic
  Interventions: Procedure: arthroscopic capsular release
- Hydro-dilatation (Active Comparator): injection of water under local anesthetic in to shoulder joint
  Interventions: Procedure: Hydro-dilatation

INTERVENTIONS:
Procedure: arthroscopic capsular release — surgical release of shoulder joint capsule
  Arms: Arthroscopic capsular release
Procedure: Hydro-dilatation — dilatation of shoulder joint capsule using water pressure under local anesthetic
  Arms: Hydro-dilatation

SUMMARY:
To compare the Oxford shoulder score at 6 months post intervention for primary frozen shoulder randomised to either an arthroscopic capsular release or hydro-dilatation

DETAILED DESCRIPTION:
All potential participants for this study will be identified by an Orthopaedic Shoulder Consultant in the shoulder clinics run at the Royal Devon and Exeter NHS trust. The patients will be screened for eligibility by a research associate (SG). The eligibility criteria will be that the patient is medically fit for an operation, and has severe primary frozen shoulder in the acute painful stage, that is deemed suitable for intervention by the consultant surgeon. The patients will be informed verbally and in writing about the trial by the research associate and informed consent will be taken.

The participating patients will be randomised in a 1:1 allocation to arthroscopic capsular release (ACR) or hydrodilatation (HD). The randomisation will be administered by a central independent randomisation service, provided by a medical secretary using a computer generated randomisation sequence, who is completely independent of the trial.

All patients will be asked to fill out a number of questionnaires prior to surgery: the Oxford Shoulder Score (OSS) and the EQ-5D. The range of movement within the shoulder joint will be documented in a standard fashion.

Each patient will then undergo the assigned procedure according to the randomisation. The ACR would be performed by one of the Consultant Shoulder surgeons in their standard manner. The Hydro-dilatation would be performed by one of the Consultant Musculoskeletal radiologists in their standard manner. This would ensure that the options at each step of the operation or procedure, such as patient positioning, approach to the shoulder joint, and the closure of the wound etc are left entirely to the discretion of the Consultant performing the procedure. This will ensure that the results of the trial can be generalised to as wide a group of patients and surgeons as possible.

After the operation, patients will be reviewed using the range of movement, OSS, a patient satisfaction score and EQ-5D at 6 weeks, 3 months, and 6 months post-operatively. A record will be kept of any complications associated with the treatment. This data will be collected with by the research associate, who is independent of either intervention.

The main analysis will investigate differences in the primary outcome measure the OSS, between the two treatment groups (ACR and HD) on an intention-to-treat basis, at 6 months post-operation. Secondary outcome measures will be analysed in a similar manner. Statistical analysis will be undertaken by a statistician blinded to the interventions. Advice will be sought from an independent statistician provided by the trust to confirm the statistical methodology.

The economic evaluation will investigate the comparative cost-effectiveness of ACR versus HD. Health outcomes within 6 months follow-up will be assessed using the EuroQoL data collected within the trial, which will be valued using the standard UK TTO tariff to produce Quality-Adjusted Life-Year (QALY) estimates.

ELIGIBILITY:
Inclusion Criteria:

* Medically fit for an operation; normal x-ray; Codmans criteria frozen shoulder

Exclusion Criteria:

* Secondary causes of frozen shoulder; rotator cuff tears found at arthroscopy or hydro-dilatation; unable to adhere to trial protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Oxford shoulder score | at 6months
  Patient reported outcome with a maximum score of 48 and minimum of 0. 48 being the best outcome. Comprises 12 questions relating to pain and function specific to the shoulder

SECONDARY OUTCOMES:
Visual analogue score | at 6 months
  pain score from 0 to 10 marked by patient on a continuous line. 0 being the worst score
clinical assessment of range of movement (external rotation, internal rotation, forward flexion and abduction) | at 6 months
  clinical assessment of range of movement using goniometer at the shoulder joint

CONTACTS AND LOCATIONS:
Overall Officials: chris smith, Principal Investigator — Royal Devon and Exeter
Locations (1):
- Royal Devon and Exeter hospital, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No